CLINICAL TRIAL: NCT02324985
Title: Phase II Study of the Effects of AP0302 5% (S-Ibuprofen Topical Gel 5%) Versus the Vehicle Control on Delayed Onset Muscle Soreness of the Elbow Flexors
Brief Title: Phase II Study of AP0302 5% Versus a Vehicle Comparator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aponia Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-005
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-01

CONDITIONS: Pain; Delayed Onset Muscle Soreness
Keywords: muscle soreness
MeSH Terms: conditions — Pain; Myalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm (Active Comparator): S-Ibuprofen Topical Gel 5%
  Interventions: Drug: S-Ibuprofen Topical Gel 5%
- Placebo Arm (Placebo Comparator): Vehicle Topical Gel
  Interventions: Drug: Vehicle Topical Gel

INTERVENTIONS:
Drug: S-Ibuprofen Topical Gel 5% — S-Ibuprofen Topical Gel 5% applied every 6 hours
  Other Names: Active Gel
  Arms: Active Arm
Drug: Vehicle Topical Gel — Vehicle Topical Gel applied every 6 hours
  Other Names: Vehicle Gel
  Arms: Placebo Arm

SUMMARY:
This study is designed to evaluate the analgesic safety and efficacy of study drug (AP0302) applied topically every 6 hours as compared to a vehicle, in subjects experiencing delayed onset muscle soreness.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of S-Ibuprofen Topical Gel 5% in reducing pain/soreness associated with delayed onset muscle soreness (DOMS).

ELIGIBILITY:
Inclusion Criteria:

* no clinically significant medical conditions
* BMI between 18-30
* negative drug, alcohol, pregnancy screens
* other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* no upper extremity workout in last 6 months
* no job requiring heavy lifting
* history of muscle disorders
* allergy or intolerance to study drug
* history of recent pain medication use
* other protocol-defined exclusion criteria may apply

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sum of pain intensity differences over 24 hours from baseline (SPID24) with movement | 0-24 hours
  SPID 24

SECONDARY OUTCOMES:
Sum of pain intensity differences over 48 hours from baseline (SPID48) with movement | 0-48 hours
  SPID 48movement
Sum of pain intensity differences over 48 hours from baseline (SPID48) at rest | 0-48 hours
  SPID 48rest

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Singla, DO, Principal Investigator — Lotus Clinical Research
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States